CLINICAL TRIAL: NCT05790395
Title: Prevention of Non-communicable Diseases Through Screening and Educating Individuals on Health-risk Behaviours in the Community
Brief Title: Prevention of NCDs Through Screening and Educating Individuals on Health-risk Behaviours in the Community
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2023-081
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Health-risk Behaviours; Non Communicable Diseases
Keywords: Health-risk Behaviours; Non Communicable Diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. The participants will receive a brief telephone intervention using the Ask, Warn, Advise, Refer and Do-it-again (AWARD) model. For the advice step, the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so.
  Interventions: Other: Theory of planned behaviour, foot-in-the-door technique, and self-determination theory intervention
- Control group (Placebo Comparator): The control group participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. However, the health ambassadors will simply advise the participants to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.
  Interventions: Other: health-risk behaviors

INTERVENTIONS:
Other: Theory of planned behaviour, foot-in-the-door technique, and self-determination theory intervention — The participants will also be asked to choose the goal that they consider easiest to achieve and encouraged to quit health-risk behaviours. The research assistant will assist in achieving the participant's health-related goals by sending WhatsApp/WeChat messages or via telephone calls once per week for the first 6 months.
  Arms: Intervention group
Other: health-risk behaviors — The participants will be simply advised to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.
  Arms: Control group

SUMMARY:
Aim: to prevent NCDs by screening and educating individuals in the community on health-risk behaviours. Specifically, we will use a mobile health and a brief self-determination theory-based intervention in helping individual change their health-risk behaviours.

Hypotheses to be tested: compared with those in the control group, the participants in the intervention group will experience significantly greater success in modifying their health-risk behaviours and will have a better health-related quality of life at 12 months follow-up.

Objectives

1. To screen individuals for health-risk behaviours and identify risk factors that may contribute to NCDs
2. To educate individuals on the importance of engaging in healthy lifestyles
3. To develop a training programme - "Train the Trainers' Toolkit", with the goal to train student nurses (Years 2 to 5) as health ambassadors to implement the project on a long-term basis.

DETAILED DESCRIPTION:
Setting:

The project will be carried out in Kwai Chung Estate, one of the largest public housing estates with many low-income families in Hong Kong.

The project consists of four phases.

Phase I:

To invite 30 university nursing students (Year 2 to 5) to become health ambassadors for the prevention of NCDs in the community.

Phase II:

To develop a training curriculum and conduct a one-day workshop for university nursing students to equip them with knowledge and skills to perform screening for individuals' health-risk behaviours and educating them to adopt healthy lifestyles.

Phase III:

To recruit 300 individuals (150 each in intervention and control groups) in Kwai Chung Estate with the aims of screening and educating health-risk behaviours and identifying risk factors that may contribute to NCDs. Activities will include putting up posters and organizing a health carnival with health education talks and health checks.

Asbury Methodist Social Service will help:

* Promotion activities (promotional posters detailing the nature and purpose of the health promotion project will be posted on notice boards at The Asbury Methodist Social Service Centres to identify potential participants)
* Provide venues for health talks and health checks for subject recruitment
* Co-organize a health carnival for subject recruitment

Phase IV:

To implement a mobile health brief intervention based on self-determination theory in helping individual change their health-risk behaviours.

Intervention:

Participants will first assess for risky behaviours using a behavioural risk factor survey. In addition, their blood pressure, body weight, height, body mass index (BMI), and health-related quality of life will be assessed.

1. Intervention group Participants will then receive a brief intervention by trained health ambassadors using the Ask, Warn, Advise, Refer and Do-it-again (AWARD) model at the time of recruitment. The brief intervention includes the following steps: (1) ask about and assess health-risk behaviours; (2) warn about the high morbidity and mortality risks associated with health-risk behaviours; (3) advise to adopt healthy lifestyle practices to benefit the health; (4) refer to hotline services on request, such as smoking cessation, alcohol treatment services and district health centres; and (5) do it again if they report failure to change a health-risk behaviour at follow-up. The health ambassadors will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so. Each participant will then receive a brief (approximately 10 minutes), individual intervention with health advice about the selected health-related lifestyle practice. The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications, including (i) 'Move Your Body', (ii) 'Eat Healthy', (iii) 'Live Alcohol Free', and (iv) 'Stay Away from Tobacco', which were developed by the Hong Kong Department of Health.

   For the first 6 months of the project period, the health ambassadors will deliver WhatsApp/WeChat messages about once per week as a reminder for the participants to adhere to their desirable health-related lifestyle practice. If a participant does not own a smartphone or is unable to receive WhatsApp/WeChat messages (uncommon in Hong Kong), the health ambassadors will make a telephone call, instead of sending a message. Participants will be assessed to determine their success in changing their targeted health-related lifestyle practice at 3, 6, and 12 months.
2. Control group The control group participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. However, the health ambassadors will simply advise the participants to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.

Subject recruitment The investigators will obtain ethical approval from the Joint CUHK-NTEC CREC. Potential participants will be assessed for eligibility, and the purpose, design, procedures, and potential benefits and risks of the study will be explained to them. Informed written consent will then be sought. All subjects will be assured that their participation will be voluntary, with no prejudice attached to refusal, and that the information they provide will be kept confidential. The researcher is responsible for its safekeeping and the only one who would have access to the raw data or study record during or after the study. After the period of storage, all raw data and records will be destroyed.

The proposed study will adhere to the Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects.

Randomization and allocation concealment Stratified block randomisation with 1:1 allocation will be conducted using varying block sizes of 2-4 to achieve an appropriate balance of participant numbers between the two groups and to optimise allocation concealment. Randomization will be performed by the research assistant, who will unseal a serially labelled, opaque envelope containing a card to indicate the group allocation. To ensure allocation concealment, the random numbers used for allocation will be computer-generated by a co-investigator before subject recruitment.

Data processing and analysis

Instruments:

A behavioural risk-factor survey will be used to collect the eligible participants' demographic and clinical data and information about their health-risk behaviours at baseline and at 3, 6, and 12 months. This questionnaire is adapted from a questionnaire used by the Hong Kong Department of Health and was used to investigate multiple health-risk behaviours among Chinese adults in Hong Kong in 2021.

The EuroQoL 5-Dimension 5-level (EQ-5D-5L) will be used to measure subjects' health-related quality of life at baseline, 6 months, and 12 months. The psychometric properties of the Chinese version of the EQ-5D-5L have been tested, and the findings indicate that this tool is a valid, reliable, and sensitive measure of health-related quality of life. A Chinese-specific EQ-5D-5L value set will enable the estimation of health utility scores applicable to the Chinese population and quality-adjusted life-years (QALY) for cost-effectiveness analysis (CEA).

SPSS for Windows (SPSS version 26.0; IBM Corp., Armonk, NY, USA) will be used for the quantitative data analysis. Descriptive statistics will be used to calculate the mean, standard deviation, and frequency of the demographic and health-risk behaviour data. The analysis including the main effect, i.e., behavioural changes at 12 months in the intervention group versus those in the control group, will be performed using a chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

Chinese adults in Kwai Chung Estate:

1. age ≥18 years
2. the presence of at least one health risk behaviour (tobacco use, harmful use of alcohol, unhealthy diet and physical inactivity)
3. able to communicate in Cantonese

Nursing students:

1. age ≥18 years
2. Year 2 to 5

Exclusion Criteria:

1. poor cognitive state or mental illness
2. participation in another related study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Abstain from health-risk behaviour | 12 months
  About 10% of participants will successfully abstain from at least one health-risk behaviour at 12-month follow-up

SECONDARY OUTCOMES:
Reduction in health-risk behaviours | 12 months
  Reduction in health-risk behaviours (≥ 50% reduction from baseline) at 12-month follow-up
Improvement in health-related quality of life | 12 months
  Improvement in health-related quality of life at 12-month follow-up compare to baseline using questionnaires
Ambassadors' knowledge and skill on providing professional health advice and support to participants about changing their health-risk behaviours | 6 months
  Improvement of ambassadors' knowledge and skill on providing professional health advice and support to participants about changing their health-risk behaviours by comparing pre-, post-training and 6-month evaluation questionnaires.
Improvement in blood pressure | 12 months
  Improvement in blood pressure at 12-month follow-up compare to baseline
Improvement in body mass index | 12 months
  Improvements in body mass index at 12-month follow-up compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Supporting Information: Study Protocol
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)